CLINICAL TRIAL: NCT04849585
Title: Evaluation of the Impact of Hospitalization in Intensive Care for COVID-19 Infection
Acronym: POSTREACOVID
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Tourcoing Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RIPH_2020_11
Record Dates: First submitted 2021-02-23; First posted 2021-04-19 (Actual); Last update posted 2022-05-10 (Actual); Status verified 2022-05

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: semi-directed entretien — semi-directed entretien

SUMMARY:
To evaluate the psychological, physical, social, professional and family impact of a hospitalization in intensive care for a covid 19 by analysis of the verbatim during a semi-structured interview.

ELIGIBILITY:
Inclusion Criteria:

* All patients hospitalized in intensive care at CH Dron for a COVID 19 who have given their agreement during their follow-up consultation

Exclusion Criteria:

* Minor patient
* Patient does not speak French
* Refusal to participate

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients hospitalized in intensive care at CH Dron for a COVID 19
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2022-06 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2023-02 (Estimated)

PRIMARY OUTCOMES:
Psychological impact of hospitalization in intensive care for a covid 19. | At day 1
  Frequency of recurring nightmares, irritability and anxious patient
Physical impact of hospitalization in intensive care for a covid 19. | At day 1
  Frequency of Handicap and resumption of professional and personal activities

CONTACTS AND LOCATIONS:
Overall Officials: Pauline THILL, MD, Principal Investigator — CH TOURCOING
Locations (1):
- CH Tourcoing, Tourcoing, France